CLINICAL TRIAL: NCT01036893
Title: The Effect of Prucalopride on the Plasma Levels of Oral Contraceptives (Ethinylestradiol and Norethisterone) in Healthy Subjects
Brief Title: M0001 Effects on Oral Contraceptive Plasma Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Movetis (Industry)
Collaborators: FOCUS GmbH (Unknown)
Responsible Party: Remi Van Den Broeck, Chief Development Officer, Movetis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M0001-C101
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral contraceptives without prucalopride (No Intervention)
- oral contraceptives with prucalopride (Active Comparator): prucalopride
  Interventions: Drug: prucalopride

INTERVENTIONS:
Drug: prucalopride — prucalopride 2 mg oral dosing o.d. for 6 days
  Arms: oral contraceptives with prucalopride

SUMMARY:
This is a randomized, open-label, two-way cross-over drug-drug interaction Phase I trial.

The objectives of this phase I trial are to investigate in healthy female subjects:

* the effect of prucalopride on the absorption of ethinylestradiol and norethisterone acetate, the active constituents of several oral contraceptives, after the first dose of prucalopride.
* the effect of multiple oral dosing of 2 mg prucalopride, for 6 days o.d. (steady state), on the pharmacokinetics of ethinylestradiol and norethisterone acetate.

This trial will be conducted in healthy females of child bearing potential, i.e. females aged between 18 and 45 years (pre-menopausal).

ELIGIBILITY:
Inclusion criteria

Subjects who meet all of the following criteria are eligible for this trial:

1. Healthy females, aged between 18 and 45 years extremes included, who have regular menstrual cycle of 28 ± 3 days for the last 6 months.
2. Adequate use of non-hormonal birth control (double-barrier method (e.g. condom and spermicide, cervical cap and spermicide) or sterilization or vasectomy of the partner or certified abstinence).
3. Subjects are not smoking for at least 6 months prior to selection.
4. A body mass index (BMI) between 18 and 27 kg/m2, extremes included.
5. The subject is in good health based on a pre-trial physical and gynaecological examination, medical history, anamnesis, electrocardiogram (ECG) and the results of biochemistry, coagulation or haematology tests or a urinalysis carried out within 4 weeks before the start of the trial. If the results of the biochemistry, coagulation or haematology tests or the urinalysis are not within the laboratory's reference ranges the subject will be included only on condition that the investigator judges that the deviations are not clinically significant.
6. Subjects voluntarily signed written Informed Consent Form (ICF) in accordance with the regional laws or regulations, prior to the first trial related activity, indicating an understanding of the purpose of this trial.
7. Subjects are willing to adhere to the treatment regimen and trial procedures described in this protocol.

Exclusion criteria

Subjects meeting any of the following criteria will be excluded from the trial:

1. History, evidence or suspicion of alcohol or drug abuse (screening and Day -1).
2. History or evidence of cardiac arrhythmias, bronchospastic or cardiovascular disease (e.g. ischemic heart disease or cerebrovascular accident), hepatic or gastrointestinal, renal or endocrine (diabetes mellitus, thyrotoxicosis), or neurological (Parkinsonism) or psychiatric, gynaecological or dermatological disease, drug allergy.
3. Clinical significant abnormal ECG-intervals of morphology of the ECG, QT >500 ms or QTcB>470 ms.
4. Use of concomitant medication or oral contraceptives within 6 weeks prior to screening, or any hormonal depot-device within 6 months prior to screening . All medication, with the exception of paracetamol should be stopped.
5. Participation in an investigational drug trial in 30 days prior to the first visit.
6. Donation of blood in the 60 days preceding the first visit.
7. Pregnancy (as confirmed by a HCG test during screening and at Day 1 of each treatment session before dosing) or breast feeding.
8. Subjects with positive results for HIV, hepatitis B or C at screening.
9. Known allergy to the trial drugs ingredients/excipients.
10. Subject has contraindications for the use of oral contraceptives (known or suspected active venous thrombo-embolic disorder, known or suspected hormone dependent malignancies, undiagnosed vaginal bleeding, coagulation disorders, menstrual cycle depending migraine, lipid metabolism disorders, hepatic disorders)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
plasma levels oral contraceptives | first days
Plasma levels oral contraceptives after steady state | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- FOCUS GmbH, Neuss, Germany

REFERENCES:
- [Derived] Van de Velde V, Vandeplassche L, Hoppenbrouwers M, Boterman M, Ausma J. Effect of prucalopride on the pharmacokinetics of oral contraceptives in healthy women. Drugs R D. 2013 Mar;13(1):43-51. doi: 10.1007/s40268-013-0008-6. PMID 23539257